CLINICAL TRIAL: NCT00570895
Title: Effect of Ascorbic Acid on Iron Absorption From Ferrous Fumarate
Brief Title: Effect of Vitamin C on Iron Absorption
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Steve Abrams, MD, Professor, Baylor College of Medicine
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: H-21063
Record Dates: First submitted 2007-12-07; First posted 2007-12-11 (Estimated); Last update posted 2020-06-26 (Actual); Status verified 2020-06

CONDITIONS: Iron Deficiency
Keywords: Iron; Absorption; Ascorbic Acid; Ferrous Fumarate
MeSH Terms: conditions — Iron Deficiencies | interventions — Ascorbic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Active Comparator): Subjects in Arm A will receive the juice without ascorbic acid in addition to the muffin with ferrous fumarate.
  Interventions: Dietary Supplement: Vitamin C
- B (Active Comparator): Subjects in Arm A will receive the juice with 25mg ascorbic acid in addition to the muffin with ferrous fumarate
  Interventions: Dietary Supplement: Vitamin C

INTERVENTIONS:
Dietary Supplement: Vitamin C — Visit 1: Subjects will receive 1mg iron-58 sulfate as an aqueous solution with 50mg ascorbic acid.
  Visit 2: Subjects will consume a meal of a bread muffin labelled with 4mg of iron-57 as ferrous fumarate, and a glass of apple juice containing 0 or 25mg ascorbic acid.
  Visit 3: During this admission the apple juice will contain either 0 or 25mg ascorbic acid, the opposite of what was given to the subject in visit 2.

SUMMARY:
Iron deficiency is a common health problem worldwide. Ferrous fumarate (a form of iron) is often added to foods in an effort to prevent iron deficiency. Vitamin C can improve the amount of iron that the body absorbs, therefore it is often added to foods too. However, we don't know if vitamin C really increases the absorption of iron from ferrous fumarate.

This study will measure the iron absorption in children from a meal containing some ferrous fumarate with and without vitamin C. The study will include 4 visits to the Children's Nutrition Research Center in Houston, TX.

DETAILED DESCRIPTION:
This study involves four outpatient visits. Two test meals will be given (during visits 2 and 3) and two blood draws will be done (visits 3 and 4). A 2-3 hour fast prior to the visit is required. Therefore, subjects may come in first thing in the morning (for breakfast meal), at lunch, or in the afternoon (snack). Subjects may be scheduled to come in during the week or on weekends; however, each individual subject will need to return at the same time of day for each subsequent visit. Visit procedures are described below.

Visit 1: Subjects will be admitted to the GCRC as an outpatient after a 2-3h fast and given a reference dose of 1mg iron-58 sulfate as an aqueous solution with 50mg ascorbic acid. They will be observed for 2h after this dose and water will be freely available. No food will be allowed. After 2h subjects will be discharged home and food allowed.

Visit 2: One to 10 days later subjects will be again admitted as an outpatient after a 2-3h fast. They will consume a meal of a bread muffin labelled with 4mg of iron-57 as ferrous fumarate, and a glass of apple juice containing 0 or 25mg ascorbic acid. The order of ascorbic acid supplementation or non-supplementation will be decided by random. No food will be allowed after the meal. After 2h subjects will be discharged home and food allowed.

Visit 3: Two weeks (+/- 3 days) later they will be readmitted after a 2-3h fast and the second visit repeated. During this admission the apple juice will contain either 0 or 25mg ascorbic acid, the opposite of what was given to the subject in visit 2. Immediately prior to administration of the second test meal, 10mL blood will be drawn for measurement of iron nutritional parameters (e.g. CBC, serum ferritin) and iron isotope ratio measurement. Incorporation of iron-57 will be used to calculate iron absorption from the test meal given during visit 2, and incorporation of iron-58 used to measure absorption from the reference dose (a measure of iron status). No food will be allowed after the meal and blood draw. After 2h subjects will be discharged home and food allowed.

Visit 4: Two weeks (+/- 3 days) later subjects will be admitted for a 10mL blood draw as described above. Incorporation of iron-57 will reflect the absorption of ferrous fumarate from the test meal given during visit 3.

ELIGIBILITY:
Inclusion Criteria:

* Healthy children
* 4-8.0y of age
* No chronic medical problems
* Not on regular medications
* Subjects on vitamin or mineral supplementation will be eligible as long as they discontinue the supplements two weeks prior to the first visit, until the end of the fourth visit.

Exclusion Criteria:

* Chronic medical problems that interfere with nutrient absorption
* History of prematurity (<37 wks gestational age)
* History of birth weight <2500g
* Current height-for-age or weight-for-age below the 5th centile or above the 95th centile

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 22 (Actual)
Dates: Start 2008-01; Primary Completion 2008-04 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Clarify the effect, if any, of ascorbic acid on ferrous fumarate absorption | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Steven A Abrams, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Children's Nutrition Research Center, Houston, Texas, United States

REFERENCES:
- [Derived] Balay KS, Hawthorne KM, Hicks PD, Griffin IJ, Chen Z, Westerman M, Abrams SA. Orange but not apple juice enhances ferrous fumarate absorption in small children. J Pediatr Gastroenterol Nutr. 2010 May;50(5):545-50. doi: 10.1097/MPG.0b013e3181b1848f. PMID 20639713